CLINICAL TRIAL: NCT02304900
Title: Effect of the Color of the Intra-eye Implant in the Cataract Surgery on the Sleep
Acronym: IOL et sommeil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRI09-PJP / IOL et sommeil
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2017-02

CONDITIONS: Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 : white implant (Experimental): Randomization will determine the color of the implant to be used for each patient for interventions in both eyes, white or yellow to know.
  Interventions: Other: white implant
- Group 2 : yellow implant (Experimental): Randomization will determine the color of the implant to be used for each patient for interventions in both eyes, white or yellow to know.
  Interventions: Other: yellow implant

INTERVENTIONS:
Other: white implant — 1. st intervention (in the month following the inclusion): Randomization of the color of the implant
  2. nd operation (1 to 3 months after the first surgery): Installation of a same color as the first implant operated eye
  Arms: Group 1 : white implant
Other: yellow implant — 1. st intervention (in the month following the inclusion): Randomization of the color of the implant
  2. nd operation (1 to 3 months after the first surgery): Installation of a same color as the first implant operated eye
  Arms: Group 2 : yellow implant

SUMMARY:
The cataract surgery (550 000 operations per year in France) is to replace the cloudy lens with a refractive implant. Two colors of implants are available: white implants, filtering out ultraviolet and yellow implants, filtering and more blue light. No clinical data are available to assert the superiority of an implant according to its color and the choice is made according to the preference of the surgeon and / or "markets".

It is established in humans that blue light has an important role on the secretion of melanopsin, a key mediator of the circadian cycle. This "clock" regulates most neuroendocrine functions in the nycthémère (sleep, mood, temperature, cortisol, ..). The question of the impact of these neuro endocrine functions of the installation of a blue light filter into the eyes of patients operated thus arises.

ELIGIBILITY:
Inclusion Criteria:

* female or male subject
* subject between 60 and 90 years old
* Visual acuteness < or = with 2 eyes
* Indication operating of the cataract

Exclusion Criteria:

* NA

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Variation between before and 2 months after surgery sleep time | 2 months

SECONDARY OUTCOMES:
Variation between before and 2 months after surgery the number of hours of sleep | 2 months
Variation between before and 2 months after surgery of the quality of sleep | 2 months
Variation between before and 2 months after surgery the mood evaluation score | 2 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service d'Ophtalmologie, Brest
  - Service d'Ophtalmologie, Centre Hospitalier Paul Martinais, Loches
  - Service d'Ophtalmologie, Tours

REFERENCES:
- [Result] Zambrowski O, Tavernier E, Souied EH, Desmidt T, Le Gouge A, Bellicaud D, Cochener B, Limousin N, Hommet C, Autret-Leca E, Pisella PJ, Camus V. Sleep and mood changes in advanced age after blue-blocking (yellow) intra ocular lens (IOLs) implantation during cataract surgical treatment: a randomized controlled trial. Aging Ment Health. 2018 Oct;22(10):1351-1356. doi: 10.1080/13607863.2017.1348482. Epub 2017 Jul 10. PMID 28691893